CLINICAL TRIAL: NCT01084343
Title: A Dose Escalating Phase I Study, Double-blind, Randomized, Placebo-controlled for Examining the Safety and Tolerability to a Prophylactic HIV-1 Vaccine Called MYM-V101, Administered i.m. in Combination With i.n. Administrations to Healthy Female Subjects.
Brief Title: Investigation of the Safety of an HIV-1 Vaccine Given Intra-muscularly and Intra-nasally to Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mymetics Corporation (Industry)
Collaborators: Kinesis Pharma B.V. (Industry); CEVAC (Unknown); M.A.R.C.O. (Unknown); Mouton's Safety Consultancy (Unknown); Pharmafour (Unknown); Pevion (Unknown); Chimera (Unknown); Institut Cochin (Other); San Raffaele University Hospital, Italy (Other); INSERM UMR 721 (Unknown)
Responsible Party: Dr. Sylvain Fleury, Mymetics Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MYM-V101-CT08-101; 2008-007306-10 (EudraCT Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2009-10

CONDITIONS: HIV-1
Keywords: vaccination; prophylaxis
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel 1 (Active Comparator): Subjects in this panel receive the low dose of vaccine (10 microgram of peptides). Twelve subjects are included in this panel, 8 of them receive the active vaccine and 4 receive the carrier only (placebo).
  Interventions: Biological: MYM-V101
- Panel 2 (Active Comparator): Subjects in this panel receive the high dose of vaccine (50 microgram of peptides). Twelve subjects are included in this panel, 8 of them receive the active vaccine and 4 receive the carrier only (placebo).
  Interventions: Biological: MYM-V101

INTERVENTIONS:
Biological: MYM-V101 — * Panel 1: 2 vaccinations in the muscles followed by 2 vaccinations in the nose, 10 microgram or placebo each, every 8 weeks.
  * Panel 2: 2 vaccinations in the muscles followed by 2 vaccinations in the nose, 50 microgram or placebo each, every 8 weeks.
  Other Names: MYM-V101.1: low dose intramuscular; MYM-V101.2: high dose intramuscular; MYM-V101.3: high dose intranasal; MYM-V101.4: low dose intranasal

SUMMARY:
This study is designed to investigate the safety and efficacy of a newly developed vaccine against HIV-1 in female healthy subjects. Safety will be assessed by local and systemic adverse reactions, investigations of blood and urine, and physical exam including vital sign measurements. Efficacy will be assessed in blood, and in vaginal and rectal mucosal samples.

DETAILED DESCRIPTION:
The current treatment of HIV is aimed at delaying the disease process after the body has been infected with the virus. HIV treatment does not prevent the spreading of the virus to uninfected people. Prevention of HIV infection could be realized by a vaccine. An effective vaccine could slow down the world wide epidemic. None of the potential vaccines investigated in the past 20 years could provide protection to HIV. All these vaccines were aimed at stimulating an immune reaction in the blood. A new theory has been raised that protection against HIV should take place at the site where the virus in most cases enters the body after sexual contacts, in the vagina and rectum. Mymetics Corporation, sponsor of this clinical trial, has developed a new vaccine, based on the so-called virosome technique. This vaccine should be able to induce a local immune reaction in the mucosa of vagina and rectum. Investigations in laboratory animals showed that the newly developed vaccine was safe and well tolerated and a local immune reaction in the mucosa could be established. The next step is to investigate if the concept of mucosal immunity does also apply in the human being. Therefore this trial is being designed to investigate if the newly developed vaccine is also safe and well tolerated in healthy subjects. In addition, it will be investigated if the vaccine can induce an immune response in the mucosa of vagina and rectum. The vaccine will be investigated for the first time in man. The vaccine consists of a very small part of the HIV 1 virus, coupled to a carrier, the virosome. The vaccine also contains two proteins of the influenza virus. These are needed for stability of the vaccine and activation of the immune system in general. There will be two groups of 12 healthy female subjects. In total 24 subjects will participate in this study. The first group will be vaccinated with a low dose of the vaccine (10 microgram of peptide). If the vaccine is assessed as safe during the safety reviews, the second group will be vaccinated with a high dose of vaccine (50 microgram of peptide). Safety and tolerability of the high dose will also be assessed during two safety reviews. Each subject will be vaccinated on four occasions, separated by eight weeks. The first two vaccinations will be given in the muscles and the third and fourth vaccination will be given in the nose in order to enhance the immune response in the mucosa. In both groups, eight subjects will be vaccinated with the real vaccine and four subjects will be vaccinated with the carrier only (placebo). Nor the investigator neither the subject will know which vaccination they receive. It will be a so-called double-blinded study. Safety and tolerability will be assessed by the local and systemic adverse reactions. In addition, blood and urine will be investigated and subjects will have a physical examination including vital signs measurements. At home, subjects will complete a diary card for the registration of local and systemic adverse events. The immune response in blood will be measured. For the investigation of the mucosal immune response, a smear from the mucosa of vagina and rectum will be taken and investigated at four visits. This will be performed with special sponges and it is a painless procedure. Total duration of the study for each subject will be 32-34 weeks. HIV infection due to this vaccination is not possible.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged between 18 and 45 years, extremes included
2. Having regular menstrual cycles (24 to 30 days). Women that got sterilized by bilateral tubal ligation are allowed, as long as they have regular cycles
3. Non-smoking or smoking (no more than 10 cigarettes or 2 cigars or 2 pipes per day, for at least 3 months prior to selection)
4. Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, extremes included. BMI is calculated as the weight (in kg) divided by the square of height (in m)
5. Informed Consent Form (ICF) signed voluntarily before first trial-related activity
6. Able to comply with all protocol requirements
7. Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, a gynecological examination, medical history, electrocardiogram, vital signs and the results of blood biochemistry and hematology tests and a urinalysis carried out at screening
8. If the subject is of childbearing potential, agrees to use adequate contraception (oral contraceptives or double barrier method, as described in section 5.2.4, point 7 of the protocol) and not become pregnant for the duration of the study.

Exclusion Criteria:

1. Male
2. Female subject without regular menstrual cycle (24-30 days)
3. History of total hysterectomy
4. Female subject of childbearing potential without use of effective birth control method(s), or not willing to continue practicing these birth control method(s) for the duration of the trial
5. Spermicides or other chemicals as used in contraceptive barrier methods (i.e., a male or female condom, diaphragm, cervical cap or intra-uterine device);
6. A positive pregnancy test or breast feeding at screening
7. A positive HIV-1 or HIV-2 test at trial screening
8. Having vaginitis as observed by local inspection and vaginal swab
9. Recurrent vaginal infections or sexually transmitted diseases within one year prior to vaccination
10. A positive test for Hepatitis A (confirmed by hepatitis A antibody IgM), hepatitis B (confirmed by hepatitis B surface antigen), or hepatitis C (confirmed by hepatitis C virus antibody) infection at trial screening
11. History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drugs which in the investigator's opinion would compromise subject safety or compliance with trial procedures
12. Currently active or underlying diabetes, gastrointestinal, cardiovascular, neurological, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, auto-immune disease(s), inheritable immune deficiency(s), infectious disease(s), nasal disorders (i.e. rhinitis, chronic nose bleeds, chronic sinusitis, polyps, chronic cold sores), dental or mouth infections, or rectal problems (fistals, hemorrhoids)
13. History of allergic disease (i.e. egg, milk, dairy products) or reaction likely to be exacerbated by any component of the vaccine to be administered in this trial, and severe allergic disease(s)
14. Contraindication to i.m. injections, history of bleeding disorder or use of anticoagulant therapy within 4 weeks prior to the first study vaccination
15. Having received any of the following substances:

    * Nasal or inhalation corticosteroids within 2 weeks prior to first vaccination
    * Vaginal and/or rectal treatment within 3 days prior to first mucosal sampling
    * HIV vaccine in a prior clinical trial
    * Immunosuppressive medications within 6 months prior to first vaccination
    * Blood products within 120 days prior to the first vaccination
    * Immunoglobulin within 60 days prior to the first vaccination
    * Any investigational or non-registered drug or vaccine within 30 days preceding the first vaccination
    * Any planned vaccination during the study period and safety follow-up
    * Allergy treatment with antigen injections, within 14 days prior to the first study vaccination
    * Current anti-tuberculosis preventive therapy or treatment
16. Serious adverse reactions to vaccines such as, but not limited to, anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain or a history of anaphylactic reactions
17. Donation of blood or plasma within the 30 days preceding the first vaccination
18. Acute disease at the time of enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Adverse events (local and systemic) | 24 weeks
  Adverse events will be collected in the CRF by the investigator. In addition, the subjects will keep a diary card in order to collect adverse events at home.

SECONDARY OUTCOMES:
Humoral immune response (in blood) | 24 weeks
  Quantification of blood antibodies (IgG and IgA).

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, Prof. Dr., Principal Investigator — CEVAC, University of Ghent, Belgium; Sylvain Fleury, PhD, Study Chair — Mymetics Corporation
Locations (1):
- CEVAC, Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels G, Maes C, Clement F, van Engelenburg F, van den Dobbelsteen M, Adler M, Amacker M, Lopalco L, Bomsel M, Chalifour A, Fleury S. Randomized Phase I: Safety, Immunogenicity and Mucosal Antiviral Activity in Young Healthy Women Vaccinated with HIV-1 Gp41 P1 Peptide on Virosomes. PLoS One. 2013;8(2):e55438. doi: 10.1371/journal.pone.0055438. Epub 2013 Feb 20. PMID 23437055
- See also: Sponsor of the trial — http://www.mymetics.com
- See also: Clinical site of the trial — http://www.cevac.be